CLINICAL TRIAL: NCT07377162
Title: HYPERMIND - Hyperoxia Effects on Cerebral Hemodynamics
Brief Title: HYPER MIND - Hyperoxia Effects on Cerebral Hemodynamics
Acronym: HYPER-MIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Fabio Taccone, MD, PHD, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SRB2023205
Record Dates: First submitted 2025-12-11; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hyperoxemia; Cerebrovascular Circulation; Cerebral Autoregulation; Critical Illness; Mechanical Ventilation
Keywords: hyperoxemia; brain hemodynamics; tcd; cerebral autoregulation; Critical Illness; intensive care unit; hyperoxia; oxygen
MeSH Terms: conditions — Critical Illness; Choroideremia; Hyperoxia

STUDY DESIGN:
Intervention Model Description: Participants will undergo one or two controlled hyperoxic stimuli depending on baseline FiO₂. All participants receive the same physiological intervention consisting of a brief increase in inspired oxygen fraction (FiO₂), with cerebral hemodynamics monitored using continuous transcranial Doppler. No randomization is performed.
Masking Description: Not applicable. This physiological study cannot be masked due to the nature of FiO₂ manipulation and continuous hemodynamic monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Hyperoxic Stimulus (Experimental): Participants receive one or two brief normobaric hyperoxic (NBHO) stimuli during mechanical ventilation. The inspired fraction of oxygen (FiO₂) is transiently increased to 0.5 or 1.0 depending on baseline FiO₂ requirements. Cerebral blood flow and autoregulation are continuously monitored using transcranial Doppler ultrasound.
  Interventions: Other: Normobaric Hyperoxic Stimulus (NBHO)

INTERVENTIONS:
Other: Normobaric Hyperoxic Stimulus (NBHO) — The intervention consists of a short, controlled increase in the inspired oxygen fraction (FiO₂) delivered by the mechanical ventilator. Depending on baseline FiO₂, patients will receive: Depending on baseline FiO₂, patients will receive:
  Two-step NBHO (baseline FiO₂ < 0.5): FiO₂ raised to 0.5 and then to 1.0 One-step NBHO (baseline FiO₂ ≥ 0.5): FiO₂ raised to 1.0 Each step includes 5 minutes to reach steady state followed by a 10-minute recording period. Cerebral blood flow velocity and autoregulation are continuously assessed using transcranial Doppler ultrasound.

SUMMARY:
This study aims to better understand how short periods of exposure to high oxygen levels affect blood flow in the brain of patients who are intubated and mechanically ventilated in the Intensive Care Unit (ICU). Many ICU patients receive more oxygen than strictly necessary, and high blood oxygen levels (hyperoxemia) are very common. However, the immediate effects of short hyperoxic exposures on cerebral circulation and autoregulation remain poorly understood.

In this study, patients who already require mechanical ventilation for medical reasons will undergo a brief and controlled increase in the oxygen delivered through the ventilator (FiO₂). During this time, we will continuously monitor blood flow in one of the main brain arteries using a non-invasive ultrasound technique called transcranial Doppler (TCD). The goal is to evaluate how cerebral blood flow, pulsatility, and autoregulatory capacity change during and after a short hyperoxic stimulus.

No additional invasive procedures are required beyond standard ICU monitoring, except for the temporary adjustment of the ventilator's oxygen settings and arterial blood gas sampling, which are part of usual care in critically ill patients. Participation does not provide direct clinical benefit but may help improve future oxygen management in ICU patients. The study involves minimal risk, as short hyperoxic exposures are already common in routine care and will be interrupted immediately in case of any adverse event.

DETAILED DESCRIPTION:
Patients will be studied under controlled mechanical ventilation with stable ventilatory, hemodynamic, and sedative settings. Continuous transcranial Doppler (TCD) monitoring will be performed using a 2-MHz probe insonating the middle cerebral artery through the temporal bone window. Cerebral blood flow velocity signals and arterial blood pressure waveforms will be recorded continuously for offline analysis.

The experimental protocol consists of stepwise increases in the fraction of inspired oxygen (FiO₂), according to baseline oxygen requirements. Patients with a baseline FiO₂ < 0.5 will undergo two consecutive hyperoxic steps (FiO₂ 0.5 followed by FiO₂ 1.0), whereas patients with a baseline FiO₂ ≥ 0.5 will undergo a single hyperoxic step (FiO₂ 1.0). Each hyperoxic step will include a stabilization period of approximately 5 minutes to allow attainment of a physiological steady state, followed by a 10-minute recording period dedicated to cerebral hemodynamic and autoregulation assessment. After completion of the hyperoxic exposure(s), FiO₂ will be returned to baseline values. In total, there will be 3 or 4 steps, depending on the baseline FiO₂.

Arterial blood gas samples will be obtained at baseline, at the end of each hyperoxic step, and after return to baseline oxygen settings to document changes in arterial oxygen and carbon dioxide tensions. Ventilation parameters, sedation, vasoactive drug infusion rates, and fluid therapy will be kept constant throughout the protocol whenever clinically feasible.

Cerebral hemodynamic assessment will include mean flow velocity, pulsatility index, and resistive index derived from TCD signals. Dynamic cerebral autoregulation will be evaluated using established indices (the mean flow index (Mxa), transfer function analysis (TFA) parameters, autoregulation index (ARI)), and metrics derived from spontaneous fluctuations in arterial blood pressure and cerebral blood flow velocity.

Analyses will primarily rely on paired statistical methods. Exploratory subgroup analyses according to baseline oxygen requirements, illness severity, or relevant comorbidities may be conducted.

Patient safety will be continuously monitored throughout the protocol, and the procedure will be immediately discontinued in case of any clinical instability, including hemodynamic deterioration, arrhythmias, or oxygenation abnormalities.

ELIGIBILITY:
Inclusion Criteria

* Adult patients aged ≥18 years
* Admitted to the intensive care unit (ICU)
* Intubated and mechanically ventilated for ≤72 hours
* Receiving volume-controlled mechanical ventilation
* Arterial partial pressure of carbon dioxide (PaCO₂) between 35 and 45 mmHg
* Invasive arterial blood pressure monitoring in place
* Adequate transcranial Doppler (TCD) acoustic window
* Clinically judged to be suitable for a brief normobaric hyperoxic stimulus
* Expected to receive one or two hyperoxic steps based on baseline FiO₂ requirements: a) Baseline FiO₂ < 0.5: two-step hyperoxic stimulus (FiO₂ 0.5 followed by FiO₂ 1.0); b) Baseline FiO₂ ≥ 0.5: one-step hyperoxic stimulus (FiO₂ 1.0)

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Extracorporeal membrane oxygenation (ECMO)
* Continuous renal replacement therapy (CRRT)
* Contraindications to hyperoxia, as judged by the treating physician
* Severe hemodynamic instability requiring changes in vasopressor dose during the recording period
* Inability to obtain a reliable transcranial Doppler signal through the temporal acoustic windows
* Any clinical condition deemed by the treating physician to pose unacceptable risk during hyperoxic exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Flow Index (Mx) During Normobaric Hyperoxia | Baseline (prior to hyperoxic exposure), during normobaric hyperoxia steps, assessed during the intervention period, and after returning to baseline (assessed up to 20 minutes)
  Dynamic cerebral autoregulation will be assessed using the mean flow index (Mx), calculated as the moving Pearson correlation coefficient between mean arterial pressure (MAP) and mean middle cerebral artery (MCA) blood flow velocity measured by transcranial Doppler ultrasonography.
  The outcome will be reported as the absolute change in Mx from baseline, calculated as the average Mx value during normobaric hyperoxia minus the baseline average.

SECONDARY OUTCOMES:
Change in Middle Cerebral Artery Cerebral Blood Flow During Normobaric Hyperoxia | Baseline (prior to hyperoxic exposure), during normobaric hyperoxia, assessed during the intervention period (up to 30 minutes per study session), and after returning to baseline (assessed up to 20 minutes)
  Cerebral hemodynamics will be assessed by transcranial Doppler ultrasonography of the middle cerebral artery (MCA). The cerebral blood flow velocity (cm/s) will be evaluated and analyzed as a change from baseline during normobaric hyperoxia. It will be expressed as the absolute change from baseline, calculated as the average value during the last 5 minutes of normobaric hyperoxia minus the baseline average.
Change in Autoregulation Index (ARI) During Normobaric Hyperoxia | Baseline (prior to hyperoxic exposure), during normobaric hyperoxia, assessed during the intervention period (up to 30 minutes per study session), and after returning to baseline (assessed up to 20 minutes)
  Cerebral autoregulation will also be evaluated using the Autoregulation Index (ARI) derived from transfer function-based step response analysis, expressed on a scale from 0 to 9. The outcome will be expressed as the absolute change from baseline during normobaric hyperoxia.
Change in Transfer Function Analysis Parameters During Normobaric Hyperoxia | Baseline (prior to hyperoxic exposure), during normobaric hyperoxia, assessed during the intervention period (up to 30 minutes per study session), and after returning to baseline (assessed up to 20 minutes)
  Transfer function analysis (TFA) between mean arterial pressure and middle cerebral artery blood flow velocity will be performed. Gain (cm/s/mmHg) will be analyzed in the low-frequency band (0.07-0.20 Hz). It will be expressed as absolute change from baseline during normobaric hyperoxia.
Change in Transfer Function Analysis Parameters During Normobaric Hyperoxia | Baseline (prior to hyperoxic exposure), during normobaric hyperoxia, assessed during the intervention period (up to 30 minutes per study session), and after returning to baseline (assessed up to 20 minutes)
  Description: Transfer function analysis (TFA) between mean arterial pressure and middle cerebral artery blood flow velocity will be performed. Phase (radians) will be analyzed in the low-frequency band (0.07-0.20 Hz). It will be expressed as absolute change from baseline during normobaric hyperoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Silvio Taccone, MD, PhD, Principal Investigator — Hôpital Erasme - Université Libre de Bruxelles (ULB)
Locations (1):
- Erasme Hospital - ULB, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the data are collected within Hôpital Erasme - ULB and contain coded clinical information that cannot be transferred outside the institution according to local ethical and data protection policies. Only aggregated, non-identifiable results will be shared through scientific publications or presentations.